CLINICAL TRIAL: NCT00691236
Title: Evaluation of Zoledronic Acid as a Single Agent and as an Adjuvant to Chemotherapy in the Management of High Grade Osteosarcoma
Brief Title: Evaluation of Zoledronic Acid as a Single Agent or as an Adjuvant to Chemotherapy in High Grade Osteosarcoma
Acronym: ZOL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Dr Manish Agarwal, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 382
Record Dates: First submitted 2008-05-27; First posted 2008-06-05 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Osteosarcoma
Keywords: osteosarcoma; zoledronic acid; bisphosphonates; adjuvant to chemotherapy
MeSH Terms: conditions — Osteosarcoma | interventions — Zoledronic Acid; Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): standard chemotherapy which is Adriamycin, Cisplatinum and Ifosfamide
  Interventions: Drug: Standard chemotherapy
- B (Experimental): zoledronic acid prior to standard chemotherapy
  Interventions: Drug: Zoledronic acid; Drug: Standard chemotherapy
- C (Experimental): zoledronic acid alone 4mg IV 3 weekly for 6 doses
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — 4mg IV 3 weekly for 6 doses
  Other Names: Zolendron,; Zometa
  Arms: B; C
Drug: Standard chemotherapy — Adriamycin + Cisplatinum and Ifosfamide
  Other Names: Doxorubicin; Holoxan
  Arms: A; B

SUMMARY:
This trial will be a pilot study to find out if zoledronic acid improves the response to chemotherapy in high grade osteosarcoma. In arm A of the study, 40 adult patients will be randomised into two groups. One group will get standard chemotherapy and the other group will get Zoledronic acid in addition to chemotherapy. The investigators will assess the histological necrosis as well as disease status for up to 2 years.

In Arm B, adult patients with relapsed disease or advanced disease who are unable to take any other therapy and are given only symptomatic care will be given 6 doses of zoledronic acid and followed up for disease status. This will be to determine the role of zoledronic acid as a single agent.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (between the ages of 18 to 65 years) with a recently diagnosed high grade osteosarcoma of the extremity
2. Non Metastatic at presentation. The metastases are ruled out by a CT scan of the chest and a PET scan.
3. Patients are willing and able to afford the standard chemotherapy.

Exclusion Criteria:

1. Non-extremity sarcomas. (pelvis and spine)
2. Age less than 18 years or greater than 65 years
3. Metastatic at presentation
4. Pregnant or lactating women
5. Renal dysfunction in the form of elevated serum creatinine
6. Dental treatment anticipated after evaluation.
7. Patients who have received or are likely to receive steroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
histological response disease free interval | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Manish Agarwal, M.S(Orth), Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India